CLINICAL TRIAL: NCT03468335
Title: Second-line Therapy With Nal-IRI After Failure Gemcitabine/Nab-paclitaxel in Advanced Pancreatic Cancer - Predictive Role of 1st-line Therapy
Brief Title: 2nd-line Therapy With Nal-IRI After Gem/Nab-pac in Advanced Pancreatic Cancer - Predictive Role of 1st-line Therapy
Acronym: PREDICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Crolll Gmbh (Other); Servier Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-PAK-0216
Record Dates: First submitted 2018-01-19; First posted 2018-03-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Second-line therapy; Nal-IRI; failure gemcitabine/nab-paclitaxel; predictive role of 1st-line therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: Open label, single arm, multicenter phase IIIb trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Cancer treatment for PDAC:
  * Nal-IRI (4.3 mg/ml) 70 mg/m2 as 1.5 hour infusion
  * 5-FU 2400 mg/m2 as 46 hour infusion
  * Folinic acid 400 mg/m2 as 0.5 hour infusion
  * all on D1 of each cycle; Cycle q2w ± 5 days
  Treatment until progressive disease or intolerable toxicity or withdrawal of consent.
  Interventions: Drug: Irinotecan Liposomal Injection [Onivyde]

INTERVENTIONS:
Drug: Irinotecan Liposomal Injection [Onivyde] — Cancer treatment for PDAC:
  * Nal-IRI (4.3 mg/ml) 70 mg/m2 as 1.5 hour infusion
  * 5-FU 2400 mg/m2 as 46 hour infusion
  * Folinic acid 400 mg/m2 as 0.5 hour infusion
  * all on D1 of each cycle; Cycle q2w ± 5 days
  Treatment until progressive disease or intolerable toxicity or withdrawal of consent.
  Other Names: Nal-IRI

SUMMARY:
Second-line therapy with Nal-IRI after failure gemcitabine/nab-paclitaxel in advanced pancreatic cancer - predictive role of 1st-line therapy

DETAILED DESCRIPTION:
Research hypothesis:

Patients profit from 2nd-line therapy with Nal-IRI if they also had a benefit from 1st-line treatment. Benefit from treatment (either 1st or 2nd-line) will be defined as a patient specific Time-To-Treatment Failure (TTF) which is in the upper third of the distribution of TTF values of the studied population.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent including participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Clinical indication for a 2nd-line systemic therapy according to current standard-of-care.
3. Age ≥ 18 years at time of study entry
4. Patients with histologically or cytologically confirmed pancreatic ductal adenocarcinoma
5. Imaging of evaluable lesions within 2 weeks of inclusion (either sonography, X-ray, CT scans, MRI)
6. ECOG performance status 0-2
7. One line of systemic gemcitabine/Nab-paclitaxel -based therapy for advanced disease (irrespective of prior adjuvant therapy) OR Previous adjuvant gemcitabine/Nab-paclitaxel-based chemotherapy with documented progression less than 6 months after termination
8. Detailed documentation of prior therapy (duration, dose-intensity, maximum toxicity, reason for discontinuation)
9. Adequate blood count, liver-enzymes, and renal function:

   * neutrophil count > 1.5 x 10^6/mL
   * Platelet count ≥ 100 x 10^9/L (≥100,000 per mm^3)
   * AST (SGOT)/ALT (SGPT) ≤ 5 x institutional upper limit of normal
   * bilirubin ≤1.5 ULN (<3 x ULN in patients with confirmed mechanical cholestasis)
   * Creatinine Clearance CLcr ≥ 30 mL/min
10. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Medical criteria:

1. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

   1. Active uncontrolled infection, chronic infectious diseases, immune deficiency syndromes
   2. Premalignant hematologic disorders, e.g. myelodysplastic syndrome
   3. Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment
   4. Prior (<3 years) or concurrent malignancy (other than biliary-tract cancer) which either progresses or requires active treatment. Exceptions are: basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a or T1b prostate carcinoma, or superficial urinary bladder tumor [Ta, Tis and T1].
   5. Pre-existing lung disease of clinical significance or with impact on performance status
   6. History or clinical evidence of CNS metastases

      Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria:

      I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of study treament. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
   7. Allogeneic transplantation requiring immunosuppressive therapy or other major immunosuppressive therapy
   8. Severe non-healing wounds, ulcers or bone fractions
   9. Evidence of bleeding diathesis or coagulopathy
   10. Major surgical procedures, except open biopsy, or significant traumatic injury within 28 days prior to star of study treatment, or anticipation of the need for major surgical procedure during the course of the study except for surgery of central intravenous line placement for chemotherapy administration.
   11. Known Gilbert-Meulengracht syndrome
   12. Known chronic hypoacusis, tinnitus or vertigo
   13. Bone marrow depression (e.g., after radiation therapy)
   14. Pernicious anemia and other megaloblastic anemias secondary to vitamin B12 deficiency
   15. Severe impairment of hepatic function
   16. Diarrhea

   Drug related criteria:
2. Medication that is known to interfere with any of the agents applied in the trial.
3. Known dihydropyrimidine dehydrogenase (DPD) deficiency
4. History of hypersensitivity to any of the study drugs or any of the constituents of the products.
5. Any other efficacious cancer treatment except protocol specified treatment at study start.

   Safety criteria:
6. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (urine or serum β-HCG acc. to SOC) at Screening.

   Methodological criteria:
7. Any experimental pretreatment for advanced disease
8. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
9. Previous enrollment in the present study (does not include screening failure).

   Regulatory and ethical criteria:
10. Patient who might be dependent on the sponsor, site or the investigator
11. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Failure of second-line treatment (TTF2) | up to 6 month
  Time-To-Treatment-Failure - (TTF2) is defined as date of signed ICF until permanent treatment discontinuation (or day of initially planned next cycle) due to progressive disease or unacceptable toxicity.
  Expected increase of the TTF2 by 50% in the cohort of patients with favorable TTF1 (TTF1 high: upper third of the patient population) as compared to patients with short TTF1 (TTF low: lowest third of the patient population)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 12 month
  Survival will be calculated from the date ICF signature until the date of death from any cause. If no event is observed (e.g. lost to follow-up) OS is censored at the day of last subject contact.
Progression Free Survival (PFS) | up to 12 month
  PFS is defined as the number of months from the date of first dose of 2nd-line treatment to the date of death or investigator assessed progression (by any imaging techique), whichever occurred earlier. If neither death nor progression is observed during the study, PFS data will be censored at the last valid tumor assessment.
AEs / SAEs | up to 12 month
  The Safety Population is the primary population for the evaluation of treatment administration/compliance and all safety data and will comprise all patients enrolled who received at least one dose of study medication. Patients will be analyzed according to the treatment actually received.
Quality of Life (QoL) EORTC QLQ-C30 | up to 6 month
  Helath related Quality of Life will be evaluated with:
  - EORTC QLQ-C30
Quality of Life (QoL) EORTC QLQ-PAN26 | up to 6 month
  Helath related Quality of Life will be evaluated with:
  - EORTC QLQ-PAN26
Quality of Life (QoL) EORTC EQ-5D-5L | up to 6 month
  Helath related Quality of Life will be evaluated with:
  - EORTC EQ-5D-5L
Evaluation of time to definitive deterioration of QoL (TDD) | from date of baseline Scrore until date QoL Score deterioration, assessed up to 12 month
  Time to QoL deterioration is defined as a loss of ≥ 10 points in the EORTC QLQ-C30 compared to base-line.
Growth modulation index (GMI) | up to 6 month
  The ratio of time to progression with the nth-line (TTP(n)) of therapy to the TTP(n-1) with the n-1th-line. GMI >1.33 is considered as a sign of activity in phase II trials.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred P. Lutz, Prof. Dr., Principal Investigator — m.lutz@caritasklinikum.de
Locations (35):
- Germany (35):
  - Klinikum St. Marien Amberg, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Hämatologisch-Onkologische Gemeinschaftspraxis, Bad Soden
  - St.Josef-Hospital Klinikum der Ruhr-Universität Bochum, Bochum
  - Städtisches Klinikum Brandenburg, Brandenburg
  - MVZ Klinikum Coburg GmbH, Coburg
  - Uniklinikum Köln GmbH, Cologne
  - Donauisar Klinikum, Deggendorf
  - BAG Onkologische Gemeinschaftspraxis Dresden, Dresden
  - MVZ Onkologische Kooperation Harz, Goslar
  - Medi Projekt, Hanover
  - Universitätsklinikum des Saarlandes, Homburg
  - DRK-Kliniken Nordhessen, Kassel
  - St. Elisabeth-Krankenhaus GmbH, Köln - Hohenlind
  - Klinikum Landshut gGmbH, Landshut
  - Onkopraxis Probstheida, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsmedizin Mannheim, Mannheim
  - Uniklinikum Marburg, Marburg
  - Krankenhaus Neuperlach, München
  - Klinikum Nürnberg Nord, Nuremberg
  - Ambulantes Therapiezentrum Hämatologie / Onkologie, Offenburg
  - Pius-Hospital, Oldenburg
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Elblandklinikum Riesa, Riesa
  - Klinikum Südstadt Rostock, Rostock
  - Caritas-Klinik St. Theresia, Saarbrücken
  - Diakonie Klinikum gGmbH, Schwäbisch Hall
  - Leopoldina Krankenhaus, Schweinfurt
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen
  - Kliniken Nordoberpfalz Klinikum Weiden, Weiden
  - Medizinische Studiengesellschaft Onkologie Nord-West GmbH, Westerstede
  - St. Josefs-Hospital, Wiesbaden
  - Hämatologisch-Onkologische Praxis Würselen, Würselen

REFERENCES:
- [Derived] Lutz MP, Ansorge N, Barmashenko G, Bauer H, Burkart C, Decker T, Ettrich T, Fischer von Weikersthal L, Geer T, Gerhardt A, Hofling S, Jacobasch L, Koenigsmann M, Leidig T, Plentz R, Rath S, Reichert D, Schulte M, Schulte N, Schwarzer A, Siegler G, Waldschmidt D, Karthaus M. Predictive criteria for overall survival and treatment duration of 2nd-line chemotherapy in patients with advanced pancreatic adenocarcinoma (AIO-PAK-0216). Br J Cancer. 2026 Jan;134(1):85-91. doi: 10.1038/s41416-025-03188-x. Epub 2025 Oct 14. PMID 41087530
- [Derived] Lahusen A, Lutz MP, Fang R, Kirchner M, Albus S, Kluck K, Karthaus M, Schwarzer A, Siegler G, Kleger A, Ettrich TJ, Becher A, Hofling S, Siveke JT, Budczies J, Tannapfel A, Stenzinger A, Cheung PF, Eiseler T, Seufferlein T. An immune responsive tumor microenvironment imprints into PBMCs and predicts outcome in advanced pancreatic cancer: lessons from the PREDICT trial. Mol Cancer. 2025 Jul 22;24(1):202. doi: 10.1186/s12943-025-02406-7. PMID 40696453